CLINICAL TRIAL: NCT04916886
Title: To Evaluate the Immunogenicity Bridging Between Different Manufacture Scales and Between Different Lots of Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) (Ad5-nCoV) in Population 6-59 Years of Age.
Brief Title: A Clinical Trial of Immunobridging and Lot-to-lot Consistency of COVID-19 Vaccine (Ad5-nCoV) in Different Age Groups.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: JSVCT118
Record Dates: First submitted 2021-05-30; First posted 2021-06-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Ad5; Immunobridging; Lot-to-lot consistency
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 50L Scale (Age 18-59) (Experimental): Single dose of 0.5ml Ad5-nCoV containing 0.5E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.5ml
- 500L Scale (Age 18-59) (Experimental): Single dose of 0.5ml Ad5-nCoV containing 0.5E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.5ml
- 800L Scale (Age 18-59) (Experimental): Single dose of 0.5ml Ad5-nCoV containing 0.5E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.5ml
- 800L Scale Lot 1 (Age 13-17) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml
- 800L Scale Lot 2 (Age 13-17) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml
- 800L Scale Lot 3 (Age 13-17) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml
- 800L Scale Lot 1 (Age 6-12) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml
- 800L Scale Lot 2 (Age 6-12) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml
- 800L Scale Lot 3 (Age 6-12) (Experimental): Single dose of 0.3ml Ad5-nCoV containing 0.3E10 vp.
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.5ml — Containing 0.5E10vp
  Arms: 500L Scale (Age 18-59); 50L Scale (Age 18-59); 800L Scale (Age 18-59)
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) 0.3ml — Containing 0.3E10vp
  Arms: 800L Scale Lot 1 (Age 13-17); 800L Scale Lot 1 (Age 6-12); 800L Scale Lot 2 (Age 13-17); 800L Scale Lot 2 (Age 6-12); 800L Scale Lot 3 (Age 13-17); 800L Scale Lot 3 (Age 6-12)

SUMMARY:
The study is a single-center, randomized and double-blinded trial to evaluate the immunobridging between different manufacture scales, lot-to-lot consistency of the Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)(Ad5-nCOV) in population 6-59 years of age. The immunobridging between different manufacture scales will be evaluated first, the immunobridging between different age groups will be evaluated second, the lot-to-lot consistency will be evaluated at last.

ELIGIBILITY:
Inclusion Criteria:

* 6-59 years of age at the time of enrollment;
* Able to provide consent or obtain consent from guardian to participate in the trial and sign an Informed Consent Form (ICF);
* Able and willing to complete all the scheduled study procedures during the whole study follow-up period;
* Axillary temperature ≤37.0℃;
* IgG ang IgM negative for Covid-19;
* Have not received any type of Covid-19 vaccines;
* No contact history of Covid-19; no travel history to medium and high risk regions and abroad in the past 21 days;
* Participants who are clinically determined to be healthy after checking medical history and physical examination are eligible to receive the product.

Exclusion Criteria:

* Medical or family history of convulsions, epilepsy, encephalopathy, and psychosis disorders;
* History of allergies to any ingredient of Ad5-nCoV, history of serious allergic reactions to any vaccine, history of allergies and immune diseases;
* Women who are pregnant or lactating, positive urine pregnancy test or plan to become pregnant during the 12 months study period;
* Acute febrile diseases and infectious diseases, medical history of SARS (SARS-CoV-1);
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and uncontrollable medications (on-site measurement for 18-59 years of age: systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg), etc;
* Severe chronic diseases or with advanced stage conditions which cannot be controlled smoothly, such as diabetes, thyroid disease, etc;
* Congenital or acquired angioedema/neurological edema;
* Urticaria history within 1 year before receiving the study vaccine;
* Asplenia or functional aspleenia;
* Thrombocytopenia or other coagulation disorders (may cause contraindications for intramuscular injection);
* Trypanophobia；
* History of receiving immunosuppressant therapy, anti-allergic therapy, cytotoxic therapy, nebulized corticosteroid therapy in the past 6 months (not including corticosteroid spray treatment for allergic rhinitis, and surface corticosteroid treatment for acute non-complicated dermatitis);
* Prior administration of blood products in last 4 months;
* Received other investigational drugs within 1 month before the study;
* Prior administration of live attenuated vaccines within 1 month before the study;
* Prior administration of subunit or inactivated vaccines within 14 days before the study;
* Current anti-tuberculosis therapy;
* Medical history of Covid-19 disease/infection;
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives or informed consent (i.e. medical, psychological, social or other conditions, etc.).

Ages: 6 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2021 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
GMT of anti SARS-CoV-2 specific neutralizing antibody | 28 days after vaccination
  GMT of anti SARS-CoV-2 specific neutralizing antibody in all groups (wild type variants test).

SECONDARY OUTCOMES:
Seroconversion rate of SARS-CoV-2 neutralizing antibody | 28 days after vaccination
  Seroconversion rate of anti SARS-CoV-2 specific neutralizing antibody (wild type variants test).
GMI of SARS-CoV-2 neutralizing antibody | 28 days after vaccination
  GMI of anti SARS-CoV-2 specific neutralizing antibody (wild type variants test).
GMT of SARS-CoV-2 S protein RBD antibody | 28 days after vaccination
  GMT of SARS-CoV-2 S protein RBD antibody measured by ELISA in all groups
Seroconversion rate of SARS-CoV-2 S protein RBD antibody | 28 days after vaccination
  Seroconversion rate of SARS-CoV-2 S protein RBD antibody measured by ELISA in all groups.
GMI of SARS-CoV-2 S protein RBD antibody | 28 days after vaccination
  GMI of SARS-CoV-2 S protein RBD antibody measured by ELISA in all groups.
GMT of Ad5 vector neutralizing antibody | 28 days after vaccination
  GMT of anti Ad5 vector neutralizing antibody responses post vaccination in all groups
GMI of Ad5 vector neutralizing antibody | 28 days after vaccination
  GMI of Ad5 vector neutralizing antibody responses post vaccination in all groups
Stratified analysis on Ad5 vector neutralizing antibody | 28 days after vaccination
  Stratified analysis based on the GMT of Ad5 vector neutralizing antibody responses post vaccination.
Incidence of Adverse Reactions/Events (AE/AR) | Within 30 minutes after vaccination
  The occurance of Adverse Reactions/Events within 30 minutes post vaccination
Incidence of Adverse Reactions/Events (AE/AR) | Within 0-7 days after vaccination
  The occurance of Adverse Reactions/Events (AE/AR) within 7 days post vaccination.
Incidence of Adverse Reactions/Events (AE/AR) | Within 0-28 days after vaccination
  The occurance of Adverse Reactions/Events (AE/AR) within 28 days post vaccination.
Incidence of Serious Adverse Events (SAE) | Within 12 months after vaccination
  Occurance of Serious Adverse Events (SAE) post vaccination.
Incidence of Adverse Events of Special Interest (AESI) | Within 12 months after vaccination
  Occurance of Adverse Events of Special Interest (AESI) post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MSD, Principal Investigator — Jiangsu Provincal Center for Disease Control and Prevention
Locations (1):
- Funing Center for Disease Control and Prevention, Yancheng, Jiangsu, China

REFERENCES:
- [Derived] Wu YF, Wei MW, Wang RJ, Guo XL, Pan HX, Gao YC, Li XL, Wang X, Ma XM, Wan P, Zhou L, Zhu YW, Li JX, Zhu FC. Immunogenicity consistency and safety with different production scales of recombinant adenovirus type-5 vectored COVID-19 vaccine in healthy adults: a randomized, double-blinded, immunobridging trial. Expert Rev Vaccines. 2023 Jan-Dec;22(1):662-670. doi: 10.1080/14760584.2023.2234997. PMID 37432025